CLINICAL TRIAL: NCT06059482
Title: The Effect of Trunk Control on Sitting Balance and Upper Extremity Functions in Patients With Subacute Stroke
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/06-10
Record Dates: First submitted 2023-07-11; First posted 2023-09-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: upper extremity; stroke; trunk control; sitting balance
MeSH Terms: conditions — Stroke | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Evaluations will be made once.

SUMMARY:
The study aims to examine whether trunk control affects sitting balance and upper extremity functions in patients with subacute stroke.

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be informed about the study and the participants who agree to participate in the study will be given the "Mini-Mental Test" and "Brunnstrom Upper Extremity Staging" tests, respectively. Then, Trunk Impairment Scale, Trunk Control Test, Function in Sitting Test, and "Fugl Meyer Upper Extremity Test" will be applied respectively.

Thirty patients with stroke will included in the study. Trunk Impairment Scale and Trunk Control Test will used to assess trunk control assessment. Fugl-Meyer Assessment of the upper extremity will used to assess upper extremity. Function in Sitting Test will used to assess sitting balance. To evaluate between correlation trunk control and upper extremity and sitting balance will used to correlation analysis tests

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with stroke and being in the subacute period (stroke onset time is between 0-6 months),
* Over 18 years old,
* Mini-Mental Test score ≥ 24 points,
* Able to sit independently in a chair for 10 minutes
* To be able to understand and follow simple explanations.

Exclusion Criteria:

* Having been diagnosed with a brain stem or cerebellar stroke,
* Having neurological or orthopedic pathology,
* Having acute low back pain,
* Having undergone surgery in the last 6 months,
* Having neglect, aphasia and heminanopsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stroke
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale | Baseline (First assessment)
  It is a scale developed for the evaluation of the trunk after stroke. It consists of 3 parts:static sitting balance, dynamic sitting balance and coordination. A maximum of 23 points can be obtained, 3 from the static section, 10 from the dynamic section, and 4 from the coordination section.
  Except for the coordination part, each part is evaluated bilaterally.
Trunk Control Test | Baseline (First assessment)
  Trunk Control Test is a test developed to evaluate trunk control. It consists of 4 parts. The test consists of the parameters of turning from the supine position to the weak and strong side, coming from the supine position to the sitting position and maintaining the sitting balance. The scoring of each section is 0-12-25. The total score is between 0-100. Higher scores indicate better trunk control of the patient.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | Baseline (First assessment)
  The Fugl-Meyer Assessment is a disease-specific impairment index designed to assess motor function, balance, sensation qualities and joint function in hemiplegic post-stroke patients.The scale consists of four categories (Shoulder/Elbow/Forearm, Wrist, Hand/Finger, and Coordination) and evaluates 23 different movements in 33 sections.The maximum score is 66 points
Function in Sitting Test (FIST) | Baseline (First assessment)
  The FIST is a clinical examination of sitting balance, designed to be conducted at the patient's bedside. Consists of 14 functional, everyday activities as test items. Each item of the test is scored between 0-4. The total score range of FIST is 0-56.

CONTACTS AND LOCATIONS:
Overall Officials: Lütfiye AKKURT, PhD, Study Director — Kutahya Health Sciences University; Güllü A YAGCIOĞLU, PhD, Study Chair — Saglik Bilimleri Universitesi; Cihan Caner AKSOY, PhD, Study Chair — Kutahya Health Sciences University; Fatıma YAMAN, MD, Study Chair — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No